CLINICAL TRIAL: NCT03850704
Title: Single Patient Use of Selinexor and Dexamethasone for a Patient With Multiple Myeloma
Status: No longer available | Type: Expanded Access
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 2019EX023
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Multiple Myeloma
Keywords: MM
MeSH Terms: conditions — Multiple Myeloma | interventions — selinexor

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Selinexor

SUMMARY:
This is an individual patient, expanded access protocol using Selinexor and dexamethasone ("Sd") for the treatment of Relapsed, Refractory multiple myeloma in a 64 year old male, "19023-UMN-01" weighing 105.7 kg. 19023-UMN-01 has IgG kappa myeloma that has relapsed after numerous treatments.

DETAILED DESCRIPTION:
Selinexor is an oral, first in class, slowly reversible, potent and Selective Inhibitor of Nuclear Export (SINE) compound that specifically blocks Exportin 1 (XPO1). It is one of the most promising investigational drugs available for this patient with clear risk and benefit assessment favoring potential benefit.

ELIGIBILITY:
Inclusion Criteria:

* Patients having relapsed/refractory multiple myeloma and neuropathy (or who are otherwise unable to tolerate bortezomib)
* Aged 18 years and older
* Patient able to provide written, informed consent to participate in and follow the KEAP Treatment Plan

Exclusion Criteria:

* Known hypersensitivity to selinexor or any excipients.
* Patient receiving any other investigational agent.
* Any concurrent uncontrolled and active medical condition or disease (e.g., uncontrolled active hypertension, uncontrolled active diabetes, active systemic infection, etc.).
* Known intolerance, hypersensitivity, or contraindication to glucocorticoids.
* Active graft versus host disease (after allogeneic stem cell transplantation).
* Active, unstable cardiovascular function:

  * Symptomatic ischemia, or uncontrolled clinically significant conduction abnormalities (e.g., patients with ventricular tachycardia on antiarrhythmics)
  * Congestive heart failure of New York Heart Association Class ≥ 3 or known leftventricular ejection fraction < 40%, or
  * Myocardial infarction within 3 months prior to C1D1.
* Significant renal impairment with ongoing dialysis treatment
* Active gastrointestinal dysfunction interfering with the patient's ability to swallow tablets, or any active gastrointestinal dysfunction that could, in the treating physician's opinion, interfere with absorption of treatment.
* Any active, serious psychiatric, medical, or other conditions/situations which, in the treating physician's opinion, could compromise the patient's safety.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Erica Warlick, MD, Principal Investigator — Division of Hematology, Oncology and Transplantation, University of Minnesota